CLINICAL TRIAL: NCT06730698
Title: Ultrasonographic Measurement of Thumb Muscle Thickness and Evaluation of Pinch and Grip Strength in First Carpometacarpal Joint Osteoarthritis: A Comparison of Early and Advanced Stages
Brief Title: Thumb Muscle Thickness and Strength in CMC Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Beylikduzu State Hospital (Other)
Responsible Party: Principal Investigator, Busra Sirin, Principle Investigator, Beylikduzu State Hospital
Other Study IDs: BeylikduzuStateH11
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early stage osteoarthritis: Early stage osteoarthritis according to Eaton-Litter classification (stage 1 and 2)
  Interventions: Other: No intervention
- Advanced stage osteoarthritis: Advanced stage osteoarthritis according to Eaton-Litter classification (stage 3 and 4)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
A total of 34 patients aged between 50-80 years, diagnosed with first carpometacarpal joint osteoarthritis based on hand radiographs taken within the last 3 months, will be included in the study from the Physical Therapy and Rehabilitation outpatient clinic. Sociodemographic data such as age, gender, height, weight, and BMI will be recorded. Based on their current radiographs, patients will be classified into two groups according to the Eaton-Littler classification: Stage 1-2 (early stage) and Stage 3-4 (advanced stage). Pain levels will be assessed using the Visual Analog Scale (VAS). Hand grip strength will be evaluated with a Jamar hand dynamometer, and pinch grip strength will be assessed with a Jamar pinch meter. The thicknesses of the abductor pollicis brevis, first dorsal interosseous, and opponens pollicis muscles will be measured using ultrasound. All assessments will be performed separately for the dominant and non-dominant hands.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50-80 years.
* Diagnosed with first carpometacarpal joint osteoarthritis.
* Presence of a hand radiograph taken within the last 3 months.
* Volunteered to participate in the study.

Exclusion Criteria:

* Refusal to participate in the study.
* Use of medications that may suppress osteoarthritis flares.
* Presence of rheumatologic diseases causing peripheral joint involvement.
* History of fractures or surgeries involving the first carpometacarpal joint.
* Presence of psychiatric disorders.
* Presence of cognitive impairments that could hinder understanding or performance of study-related tasks.

Ages: 50 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population includes patients aged 50-80 years with first carpometacarpal joint osteoarthritis, classified into early and advanced stages based on radiographs, excluding those with confounding medical or cognitive conditions.
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Thumb Muscle Thickness (Ultrasound) | 0 day
  Measurement of the thickness of three thumb muscles-abductor pollicis brevis, first dorsal interosseous, and opponens pollicis-using ultrasonography. These measurements will help determine muscle atrophy or hypertrophy related to disease severity and stage

SECONDARY OUTCOMES:
Grip Strength | 0 day
  Assessed using a Jamar hand dynamometer. This measure evaluates overall hand strength, which is often impaired in advanced stages of carpometacarpal joint osteoarthritis.
Pinch Strength | 0 day
  Assessed using a Jamar pinch meter. This measure evaluates the strength of the thumb-index finger pinch, a critical function for fine motor activities. It is particularly relevant to functional limitations seen in osteoarthritis.
Pain Level (VAS) | 0 day
  Pain intensity will be measured using the Visual Analog Scale (VAS). Patients will mark their perceived pain level on a 10 cm scale, providing a quantitative measure of pain severity in both early and advanced stages.

CONTACTS AND LOCATIONS:
Overall Officials: Büşra Şirin Ahısha, Principal Investigator — Beylikdüzü State Hospital
Locations (1):
- Beylikdüzü State Hospital, Istanbul, Beylikdüzü, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No